CLINICAL TRIAL: NCT00004003
Title: A Study of Gemcitabine, Cisplatin, and 5-Fluorouracil in the Treatment of Advanced Pancreatic Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Stage III or Stage IV Pancreatic Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067213; P30CA022453 (NIH); WSU-D-1993; WSU-04-03-99-M01-FB; NCI-G99-1553
Record Dates: First submitted 1999-11-01; First posted 2004-02-12 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cisplatin; Fluorouracil; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating adult patients who have stage III or stage IV pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the overall survival in patients with unresectable stage III or IV pancreatic adenocarcinoma treated with gemcitabine, cisplatin, and fluorouracil. II. Determine the resectability rate with curative intent in patients with unresectable stage III pancreatic adenocarcinoma treated with this regimen. III. Assess the tolerability and toxicity of this treatment regimen in this patient population. IV. Evaluate this regimen in terms of response rate, response duration, and overall time to disease progression in these patients. V. Evaluate the quality of life in these patients.

OUTLINE: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15, followed by cisplatin IV over 30 minutes on days 1 and 15. Patients receive fluorouracil as a continuous infusion on days 1-15. Courses repeat every 28 days. Quality of life is assessed every 28 days.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed pancreatic adenocarcinoma Unresectable locally advanced (stage III) OR Metastatic (stage IV) Gallbladder or biliary tract cancer allowed No endocrine tumors or lymphoma of the pancreas No CNS metastases

PATIENT CHARACTERISTICS: Age: Adult Performance status: SWOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL AST no greater than 3.0 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Other: No active infection No other serious systemic disorders No other active malignancies within the past year except curatively treated basal cell skin cancer or carcinoma in situ of the cervix Must have central venous access device (i.e., Infusaport or PASPORT) Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for locally advanced or metastatic disease At least 6 months since prior adjuvant chemotherapy No prior gemcitabine Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1999-04; Primary Completion 2001-11 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Philip, MD, PhD, FRCP, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States